CLINICAL TRIAL: NCT01924767
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of 4 Multiple Rising Oral Doses (2.5 mg to 100 mg) of BI 10773 Tablets in Male and Female Type 2 Diabetic Patients
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Doses of BI 10773 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.2; 2007-000654-32 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-08-09; First posted 2013-08-16 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

ARMS (4):
- BI 10773 (dose group 3) (Experimental): multiple doses as tablet
  Interventions: Drug: BI 10773 Placebo; Drug: BI 10773
- BI 10773 (dose group 4) (Experimental): multiple doses as tablet
  Interventions: Drug: BI 10773; Drug: BI 10773 Placebo
- BI 10773 (dose group 1) (Experimental): multiple doses as tablet
  Interventions: Drug: BI 10773 Placebo; Drug: BI 10773
- BI 10773 (dose group 2) (Experimental): multiple doses as tablet
  Interventions: Drug: BI 10773 Placebo; Drug: BI 10773

INTERVENTIONS:
Drug: BI 10773 Placebo — po taken fasting with 240 mL water
  Arms: BI 10773 (dose group 2)
Drug: BI 10773 — po taken fasting with 240 mL water
  Arms: BI 10773 (dose group 4)
Drug: BI 10773 Placebo — po taken fasting with 240 mL water
  Arms: BI 10773 (dose group 3)
Drug: BI 10773 — po taken fasting with 240 mL water
  Arms: BI 10773 (dose group 3)
Drug: BI 10773 Placebo — po taken fasting with 240 mL water
  Arms: BI 10773 (dose group 1)
Drug: BI 10773 Placebo — po taken fasting with 240 mL water
  Arms: BI 10773 (dose group 4)
Drug: BI 10773 — po taken fasting with 240 mL water
  Arms: BI 10773 (dose group 2)
Drug: BI 10773 — po taken fasting with 240 mL water
  Arms: BI 10773 (dose group 1)

SUMMARY:
To investigate safety, tolerability, pharmacokinetics and pharmacodynamics of BI 10773 with repeat dosing for eight days and the exploration of the pharmacokinetics and pharmacodynamics of BI 10773 after multiple dosing, including dose proportionality and assessment of steady state.

ELIGIBILITY:
Inclusion criteria:

1. Male and postmenopausal or hysterectomised female patients with proven diagnosis of type 2 diabetes mellitus treated with diet and exercise only or on a maximum of two oral antidiabetic agents except thiazolidindiones with at least one agent taken at 50% of its maximum dose or less.
2. Glycosylated haemoglobin A1 (HbA1c) £ 8.5 % at screening.
3. Age >21 and Age <70 years (male and hysterectomised female patients) Age >60 and Age <70 years (postmenopausal female patients)
4. Body Mass Index (BMI) >18.5 and <40 kg/m2
5. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion criteria:

1. Antidiabetic treatment with insulin or glitazones or with more than one oral hypoglycaemic agent (except if 2 agents and at least one of them not taken at more than 50% of its maximum dose)
2. Fasted blood glucose > 240 mg/dl (>13.3 mmol/L) on two consecutive days during washout.
3. Glycosylated haemoglobin A1 (HbA1c) >8.5% at screening
4. Clinically relevant concomitant diseases other than type 2 diabetes, hyperlipidaemia and medically treated hypertension, such as:

   * Any late stage complication of diabetes (e.g. retinopathy, polyneuropathy, vegetative disorders, diabetic foot)
   * Renal insufficiency (calculated creatinine clearance < 80 ml/min/1.73m²)
   * Cardiac insufficiency NYHA II-IV, myocardial infarction, other known cardiovascular diseases including hypertension > 160/95mmHg (measured at training visit and each of the timepoints of Day -1), stroke and TIA (Transistoric ischaemic attack)
   * Neurological disorders (such as epilepsy) or psychiatric disorders
   * Acute or relevant chronic infections (e.g. HIV, repeated urogenital infections)
   * Any gastrointestinal, hepatic, respiratory, endocrine or immunological disorder
5. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
6. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
7. A history of additional risk factors for TdP (torsade des pointes) (e.g., heart failure, hypokalemia, family history of sudden death before the age of 50)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-07; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1245.2.1 Boehringer Ingelheim Investigational Site, Neuss, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase I trial was randomised, double-blind, and placebo-controlled within dose groups. It was to be performed in 48 female and male patients with type 2 diabetes in 4 sequential groups of 12 patients each. Within each dose group, 9 patients were to receive active drug and 3 were to receive placebo.
Pre-assignment Details: 14 days wash-out of previous antidiabetic therapy followed by 8 days of once daily dosing at each dose level.
Groups:
- Placebo: Patients were treated with matching placebo as tablet once daily (qd) in the morning.
- Empagliflozin 2.5 mg qd: Patients were treated with 2.5 mg Empagliflozin as tablet once daily (qd) in the morning.
- Empagliflozin 10 mg qd: Patients were treated with 10 mg Empagliflozin as tablet once daily (qd) in the morning.
- Empagliflozin 25 mg qd: Patients were treated with 25 mg Empagliflozin as tablet once daily (qd) in the morning.
- Empagliflozin 100 mg qd: Patients were treated with 100 mg Empagliflozin as tablet once daily (qd) in the morning.
Period: Overall Study
Arm/Group | Placebo | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Started | 12 | 9 | 9 | 9 | 9
Completed | 11 | 9 | 8 | 9 | 9
Not Completed | 1 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set includes all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Placebo: Patients were treated with matching placebo as tablet once daily in the morning.
- Empagliflozin 2.5 mg qd: Patients were treated with 2.5 mg Empagliflozin as tablet once daily in the morning.
- Empagliflozin 10 mg qd: Patients were treated with 10 mg Empagliflozin as tablet once daily in the morning.
- Empagliflozin 25 mg qd: Patients were treated with 25 mg Empagliflozin as tablet once daily in the morning.
- Empagliflozin 100 mg qd: Patients were treated with 100 mg Empagliflozin as tablet once daily in the morning.
- Total: Total of all reporting groups
Arm/Group | Placebo | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd | Total
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (6.4) | 53.9 (10.9) | 51.8 (10.7) | 58.9 (8.8) | 60.3 (5.6) | 56.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 2 | 2 | 9
  Male | 10 | 7 | 8 | 7 | 7 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinically Relevant Findings in Physical Examination, Vital Signs and Clinical Laboratory Tests
Description: Percentage of participants with clinically relevant findings in physical examination, vital signs and clinical laboratory tests. Relevant findings or worsenings of baseline conditions were reported as Adverse Events (cardiac disorders and investigations).
Time Frame: day 1 to day 21
Population: Treated set.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9
percentage of participants
  Cardiac disorders | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Investigations: Hepatic enzyme increased | 8.3 | 0.0 | 0.0 | 0.0 | 0.0

2. Primary Outcome: Percentage of Participants With Clinically Relevant Findings in Electrocardiogram (ECG) Results
Description: Percentage of participants with clinically relevant findings in electrocardiogram (ECG) results
Time Frame: day 1 to day 21
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9
percentage of participants
  Clinically relevant | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Clinically irrelevant | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

3. Primary Outcome: Micturition Frequency
Description: Micturition frequency is reported as change from pre-treatment to day 9 during the day, the night and total. Baseline is the mean of days 8-3 before drug administration.
Time Frame: Baseline and Day 9
Population: Treated set
Measure: Mean (Standard Deviation); unit: frequency of micturition
Arm/Group | Placebo | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9
frequency of micturition
  Micturition day frequency | 4.1 (1.8) | 2.6 (2.1) | 5.0 (1.6) | 3.9 (1.5) | 4.4 (2.1)
  Micturition night frequency | 0.3 (1.6) | 0.2 (1.2) | 0.5 (0.5) | 0.6 (1.6) | 0.7 (0.9)
  Micturition total frequency | 4.5 (2.1) | 2.8 (2.6) | 5.5 (1.5) | 4.4 (2.4) | 5.1 (2.2)

4. Primary Outcome: Assessment of Tolerability by Investigator
Description: Tolerability will be assessed by the investigator according to the categories good, satisfactory, not satisfactory and bad.
Time Frame: day 21
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9
percentage of participants
  Good | 91.7 | 100.0 | 100.0 | 100.0 | 100.0
  Satisfactory | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Not satisfactory | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Bad | 8.3 | 0.0 | 0.0 | 0.0 | 0.0

5. Secondary Outcome: Concentration of the Analyte in Plasma
Description: Maximum concentration of the analyte in plasma (Cmax) after first dose, Maximum, minimum (Cmin) and average (Cavg) concentration of the analyte in plasma at steady-state, Concentration of analyte in plasma at 24 h after administration of the 8th dose (at steady-state) (C24,8)
Time Frame: -0:05 before dose and 0:10,0:20,0:30,0:40,1h,1:30h,2h,3h,4h,6h,8h,12h,16h,24h,30h,36h and 48h after dose on day 1.-0:05 before dose and 0:10,0:20,0:30,0:40,1h,1:30h,2h,3h,4h,6h,8h,12h,16h,24h,30h,36h, 48h,60h and 72h after dose on day 9.
Population: Pharmacokinetic set (PK set) contains of all patients who received study medication and have evaluable pharmacokinetic parameter data. The PK set will not contain placebo patients.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 9 | 9 | 9 | 9
nmol/L
  Cmax after first dose | 61.3 (20.5) | 240 (21.2) | 592 (23.7) | 2670 (26.1)
  Cmax at steady-state (N=9,8,9,8) | 66.6 (26.7) | 272 (30.1) | 622 (17.4) | 2700 (20.9)
  Cmin at steady-state (N=9,8,9,8) | 4.41 (36.9) | 23.5 (31.5) | 47.1 (35.3) | 243 (32.0)
  Cavg at steady-state (N=9,8,9,8) | 19.2 (24.3) | 83.5 (17.4) | 204 (21.5) | 922 (28.7)
  C24,8 (N=9,8,9,8) | 4.55 (36.8) | 23.8 (31.7) | 47.2 (35.2) | 249 (27.6)
Statistical Analysis 1: Comparison: Empagliflozin 2.5 mg qd vs Empagliflozin 100 mg qd; This was non-confirmatory testing, dose proportionality of dose from 2.5mg to 100mg for Cmax (single dose) was analysed; Test type: Superiority or Other; Regression, Linear; Geometric Mean of ratio = 43.661, 95% CI 2-sided [27.520 to 69.269]
Statistical Analysis 2: Comparison: Empagliflozin 2.5 mg qd vs Empagliflozin 100 mg qd; This was non-confirmatory testing, dose proportionality of dose from 2.5mg to 100mg for Cmax,ss (Multiple dose) was analysed; Test type: Superiority or Other; Regression, Linear; Geometric Mean of ratio = 31.234, 95% CI 2-sided [12.193 to 80.011]

6. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval (AUC)
Description: AUC0-∞: from 0 extrapolated to infinity after first dose AUCtau,1: over a uniform dosing interval tau after first dose AUCtau,ss: over a uniform dosing interval tau at steady-state AUCs were computed using the linear up/log down algorithm. If an analyte concentration was equal to or higher than the preceding concentration, the linear trapezoidal method was to be used. If the analyte concentration was smaller than the preceding concentration, the logarithmic method was to be used.
Time Frame: as for outcome 5
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 9 | 9 | 9 | 9
nmol*h/L
  AUC0-∞ after first dose | 468 (19.6) | 1890 (14.7) | 4780 (23.7) | 23300 (19.4)
  AUC0-24 after first dose | 397 (17.6) | 1620 (13.5) | 4200 (23.6) | 19700 (17.6)
  AUC0-tau at steady state (N=9,8,9,8) | 460 (24.3) | 2000 (17.4) | 4890 (21.5) | 22100 (28.7)
Statistical Analysis 1: Comparison: Empagliflozin 2.5 mg qd vs Empagliflozin 100 mg qd; This was non-confirmatory testing, dose proportionality of dose from 2.5mg to 100mg for AUC (0-infinity, single dose) was analysed; Test type: Superiority or Other; Regression, Linear; Geometric mean of ratio = 49.707, 95% CI 2-sided [33.490 to 73.776]
Statistical Analysis 2: Comparison: Empagliflozin 2.5 mg qd vs Empagliflozin 100 mg qd; This was non confirmatory testing, dose proportionality of dose from 2.5mg to 100mg for AUC (0-infinity, at steady state, day 9) was analysed; Test type: Superiority or Other; Regression, Linear; Geometric mean of ratio = 37.632, 95% CI 2-sided [15.429 to 91.789]

7. Secondary Outcome: Time to Maximum Concentration of the Analyte in Plasma
Description: Time from last dosing to maximum concentration of the analyte in plasma (tmax) after first dose and at steady-state
Time Frame: as for outcome 5
Population: PK set
Measure: Median (Full Range); unit: h
Arm/Group | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 9 | 9 | 9 | 9
h
  tmax after first dose | 1.50 (27.5) [0.667 to 1.50] | 1.50 (18.2) [0.983 to 2.00] | 1.50 (38.5) [0.983 to 4.00] | 3.00 (77.8) [0.983 to 4.00]
  tmax at steady-state (N=9,8,9,8) | 1.50 (27.4) [0.983 to 2.00] | 1.50 (24.3) [0.983 to 2.00] | 2.00 (62.6) [0.667 to 4.20] | 1.50 (62.3) [0.983 to 4.00]

8. Secondary Outcome: Terminal Rate Constant in Plasma
Description: Terminal rate constant in plasma after first dose and at steady-state
Time Frame: -0:05 before dose and 0:10,0:20,0:30,0:40,1h,1:30h,2h,3h,4h,6h,8h,12h,16h,24h,30h,36h and 48h after dose on day 1. -0:05 before dose and 0:10,0:20,0:30,0:40,1h,1:30h,2h,3h,4h,6h,8h,12h,16h,24h,30h,36h, 48h,60h and 72h after dose on day 9.
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 9 | 9 | 9 | 9
1/h
  Terminal rate after first dose | 0.0618 (22.4) | 0.0586 (11.5) | 0.0654 (19.9) | 0.0527 (26.8)
  Terminal rate at steady-state (N=9,8,9,8) | 0.0686 (18.5) | 0.0491 (17.5) | 0.0658 (18.8) | 0.0409 (48.4)

9. Secondary Outcome: Half-life and Mean Residence Time of the Analyte in Plasma
Description: Terminal half life of the analyte in plasma (t1/2) and mean residence time of the analyte in the body after single oral administration (MRTpo) after first dose and at steady-state.
Time Frame: as for outcome 8
Population: PK Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 9 | 9 | 9 | 9
h
  t1/2 after first dose | 11.2 (22.4) | 11.8 (11.5) | 10.6 (19.9) | 13.2 (26.8)
  t1/2 at steady state (N=9,8,9,8) | 10.1 (18.5) | 14.1 (17.5) | 10.5 (18.8) | 17.0 (48.4)
  MRT po after first dose | 12.2 (12.4) | 12.1 (19.1) | 11.0 (13.5) | 12.7 (19.7)
  MRT po at steady-state (9,8,9,8) | 10.7 (14.2) | 13.5 (22.7) | 11.2 (13.7) | 14.6 (20.6)

10. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase
Description: Apparent volume of distribution during the terminal phase (Vz/F) after first dose and at steady state. Apparent volume is defined as CL/F divided by the terminal rate constant in plasma (either after first dose or at steady-state).
Time Frame: as for outcome 8
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 9 | 9 | 9 | 9
L
  Vz/F after first dose | 192 (27.2) | 200 (19.5) | 177 (27.9) | 181 (35.1)
  Vz/F at steady state (N=9,8,9,8) | 176 (25.0) | 225 (25.9) | 172 (21.7) | 245 (56.7)

11. Secondary Outcome: Amount of Analyte Eliminated in Urine
Description: Amount of analyte that is eliminated in urine after first dose and at steady state from the time interval 0 to 24 h (Ae0-24) and 0 to 48 h (Ae0-48)
Time Frame: 0-2, 2-4, 4-6, 6-8, 8-12, 12-16, 16-24, 24-36, 36-48 hours (h) after dose on day 1 and 0-2, 2-4, 4-6, 6-8, 8-12, 12-16, 16-24, 24-36, 36-48 and 48-72 hours (h) after dose on day 9
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol
Arm/Group | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 9 | 9 | 9 | 9
nmol
  Ae0-48 after first dose | 706 (24.7) | 2570 (42.2) | 5250 (52.0) | 18500 (32.7)
  Ae0-48 at steady-state (N=9,8,8,9) | 941 (32.1) | 4530 (23.5) | 8450 (42.7) | 22400 (145)
  Ae0-24 after first dose | 613 (26.9) | 2250 (42.7) | 4770 (54.6) | 16600 (34.3)
  Ae0-24 at steady-state (N=9,8,8,9) | 820 (33.9) | 4040 (26.7) | 7520 (43.6) | 19300 (153)

12. Secondary Outcome: Fraction of Analyte Excreted Unchanged in Urine
Description: Fraction of analyte excreted unchanged in urine in the time interval 0 to 12 h (fe0-12) after first dose and at steady-state. The fraction excreted was calculated by dividing Ae0-12 by the Dose and multiply it with 100.
  Fraction of analyte excreted unchanged in urine in the time interval 0 to 24 h (fe0-24) after first dose and at steady-state. The fraction excreted was calculated by dividing Ae0-24 by the Dose and multiply it with 100.
Time Frame: as for outcome 11
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent of analyte
Arm/Group | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 9 | 9 | 9 | 9
percent of analyte
  fe0-12 after first dose | 8.50 (31.9) | 8.43 (39.8) | 6.30 (78.2) | 6.17 (37.6)
  fe0-12 at steady-state (N=9,8,8,9) | 10.6 (47.0) | 14.7 (26.5) | 9.22 (54.0) | 6.68 (154)
  fe0-24 after first dose | 11.1 (26.9) | 10.1 (42.7) | 7.38 (73.0) | 7.48 (34.3)
  fe0-24 at steady-state (N=9,8,8,9) | 14.8 (33.9) | 18.2 (26.7) | 11.4 (53.6) | 8.71 (153)

13. Secondary Outcome: Apparent and Renal Clearance of the Analyte in Plasma
Description: Apparent clearance of the analyte in plasma (CL/F) after first dose and at steady-state, Renal clearance of the analyte in plasma after extravascular administration (CLR) after first dose and at steady-state.
  Apparent clearance after first dose is defined as the dose divided by AUC0-∞; apparent clearance at steady-state is defined as the dose divided by AUC0-tau at steady-state.
  Renal clearance CLR(0-t) is defined as Ae0-t divided by AUC0-t.
Time Frame: as for outcome 8
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 9 | 9 | 9 | 9
mL/min
  CL/F after first dose | 198 (19.6) | 195 (14.7) | 193 (23.7) | 159 (19.4)
  CL/F at steady-state (N=9,8,9,8) | 201 (24.3) | 184 (17.4) | 189 (21.5) | 167 (28.7)
  CLR (0-48h) after first dose | 26.7 (42.9) | 23.5 (33.0) | 18.8 (53.1) | 13.9 (44.1)
  CLR (0-24h) at steady-state (N=9,8,8,9) | 29.7 (52.0) | 33.6 (24.9) | 21.7 (47.1) | 22.2 (83.3)

14. Secondary Outcome: Peak Trough Fluctuation
Description: Peak trough fluctuation (PTF) is defined as the difference between Cmax and Cmin divided by Cavg and multiplied with 100% at steady-state
Time Frame: as for outcome 8
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: PTF(%) of Empagliflozin
Arm/Group | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 9 | 8 | 9 | 8
PTF(%) of Empagliflozin | 323 (20.6) | 294 (28.4) | 281 (26.4) | 265 (31.9)

15. Secondary Outcome: Linearity Index
Description: The linearity index is defined as AUC0-tau divided by AUC0-∞ both at steady state.
Time Frame: as for outcome 8
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fraction
Arm/Group | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 9 | 8 | 9 | 8
Fraction | 0.983 (8.42) | 1.05 (2.39) | 1.02 (11.4) | 0.962 (19.7)

16. Secondary Outcome: Accumulation Ratios
Description: Accumulation ratio based on Cmax (RA,Cmax) and Accumulated ratio based on AUC0-tau (RA,AUC) at steady-state.
  Accumulation ratio for the respective doses were calculated using below mentioned equations:
  RA,Cmax = Cmax,ss/Cmax
  RA,AUC= AUCtau,ss/AUCtau
Time Frame: as for outcome 8
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 9 | 8 | 9 | 8
Ratio
  Accumulation ratio based on Cmax | 1.09 (27.0) | 1.13 (20.9) | 1.05 (22.3) | 0.972 (36.8)
  Accumulated ratio based on AUC0-tau | 1.16 (8.39) | 1.23 (6.17) | 1.16 (11.9) | 1.12 (20.7)

17. Secondary Outcome: Change From Baseline to Day 8 in Urinary Glucose Excretion
Description: Change from baseline to day 8 in urinary glucose excretion. Baseline is defined as Day -2.
Time Frame: -2-0 hours(h) before drug administration and 0-2, 2-4, 4-6, 6-8, 8-12,12-16 and 16-24 h after drug administration on day -2 and day 8
Population: Pharmacodynamic (PD) analysis set (PDS) contains of all patients who received study medication and have evaluable pharmacodynamic parameter data.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Placebo | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 11 | 9 | 8 | 9 | 9
mg | -3254.43 (8250.43) | 34638.37 (16226.22) | 78709.87 (53463.52) | 74030.40 (35378.01) | 88040.32 (20265.87)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 2.5 mg qd; The mean change from baseline (day -2) to day 8 and comparisons to placebo for Urine Glucose Excretion (AE(0-24)); Test type: Superiority or Other; p = 0.0067, ANCOVA — This was non-confirmatory testing; The baseline value has been used a continuous covariate; Mean Difference (Final Values) = 37645.43, 95% CI 2-sided [11021.57 to 64269.30]
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 10 mg qd; The mean change from baseline (day -2) to day 8 and comparisons to placebo for Urine Glucose Excretion (AE(0-24)); Test type: Superiority or Other; p < 0.0001, ANCOVA — This was non-confirmatory testing; The baseline value has been used a continuous covariate; Mean Difference (Final Values) = 82898.20, 95% CI 2-sided [55344.83 to 110451.6] — Mean difference to placebo is calculated
Statistical Analysis 3: Comparison: Placebo vs Empagliflozin 25 mg qd; The mean change from baseline (day -2) to day 8 and comparisons to placebo for Urine Glucose Excretion (AE(0-24)); Test type: Superiority or Other; p < 0.0001, ANCOVA — This was non-confirmatory testing; The baseline value has been used a continuous covariate; Mean Difference (Final Values) = 79982.89, 95% CI 2-sided [53087.22 to 106878.6] — Mean Difference to placebo is calculated
Statistical Analysis 4: Comparison: Placebo vs Empagliflozin 100 mg qd; The mean change from baseline (day -2) to day 8 and comparisons to placebo for Urine Glucose Excretion (AE(0-24)); Test type: Superiority or Other; p < 0.0001, ANCOVA — This was non-confirmatory testing; The baseline value has been used a continuous covariate; Mean Difference (Final Values) = 91306.96, 95% CI 2-sided [64685.41 to 117928.5] — Mean Difference to placebo was calculated

18. Secondary Outcome: Mean Daily Glucose
Description: Change from baseline to Day 8 in mean daily glucose. Baseline is defined as Day -2.
Time Frame: 0:00, 2:00, 5:00, 7:00, 10:00, 12:00,13:30 and 24:00 hours(h) after drug administration on day -2 and -0.05, 2:30, 5:00, 7:00, 10:00, 12.00, 13:30 and 24:00 hours (h) after drug administration on day 8
Population: PDS
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 11 | 9 | 8 | 9 | 9
mg/dL | -13.85 (21.39) | -27.03 (24.59) | -34.04 (19.43) | -25.89 (18.00) | -30.96 (25.03)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 2.5 mg qd; The mean percent decrease in Mean daily glucose from baseline with treatment compared with placebo from baseline -2 to day 8; Test type: Superiority or Other; p = 0.0449, ANCOVA — This was non-confirmatory testing; The baseline value has been used a continuous covariate; Mean Difference (Final Values) = -15.456, 95% CI 2-sided [-30.543 to -0.369] — Mean difference to placebo was calculated
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 10 mg qd; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.0042, ANCOVA — This was non-confirmatory testing; The baseline value has been used a continuous covariate; Mean Difference (Final Values) = -23.467, 95% CI 2-sided [-39.085 to -7.848] — Mean difference to placebo was calculated
Statistical Analysis 3: Comparison: Placebo vs Empagliflozin 25 mg qd; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.0521, ANCOVA — This was non-confirmatory testing; The baseline value has been used a continuous covariate; Mean Difference (Final Values) = -14.956, 95% CI 2-sided [-30.057 to 0.145] — Mean difference to placebo was calculated
Statistical Analysis 4: Comparison: Placebo vs Empagliflozin 100 mg qd; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.1676, ANCOVA — This was non-confirmatory testing; The baseline value has been used a continuous covariate; Difference to placebo = -10.602, 95% CI 2-sided [-25.848 to 4.644] — Mean difference to placebo was calculated

19. Secondary Outcome: Fasting Plasma Glucose
Description: Percentage change from baseline to Day 8 in fasting plasma glucose. Baseline is defined as Day -2.
Time Frame: -0:30 (Pre dose samples)
Population: PDS
Measure: Mean (Standard Deviation); unit: percentage of fasting plasma glucose
Arm/Group | Placebo | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 11 | 9 | 8 | 9 | 9
percentage of fasting plasma glucose | -15.88 (12.88) | -21.01 (6.38) | -25.69 (9.88) | -14.21 (26.00) | -24.85 (8.18)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 2.5 mg qd; The mean percent change in Fasting Plasma Glucose from baseline with treatment compared with placebo from baseline -2 to day 8; Test type: Superiority or Other; p = 0.2239, ANCOVA — This was non-confirmatory testing; The baseline value has been used a continuous covariate; Mean Difference (Final Values) = -7.269, 95% CI 2-sided [-19.162 to 4.624] — Mean difference to placebo was calculated
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 10 mg qd; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.0421, ANCOVA — This was non-confirmatory testing; The baseline value has been used a continuous covariate; Mean Difference (Final Values) = -12.844, 95% CI [-25.205 to -0.484] — Mean difference to placebo was calculated
Statistical Analysis 3: Comparison: Placebo vs Empagliflozin 25 mg qd; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.6527, ANCOVA — This was non-confirmatory testing; The baseline value has been used a continuous covariate; Mean Difference (Final Values) = -2.719, 95% CI 2-sided [-14.842 to 9.403] — Mean difference to placebo was calculated
Statistical Analysis 4: Comparison: Placebo vs Empagliflozin 100 mg qd; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.1318, ANCOVA — This was non-confirmatory testing; The baseline value has been used a continuous covariate; Mean Difference (Final Values) = -8.998, 95% CI 2-sided [-20.818 to 2.822] — Mean difference to placebo was calculated

20. Secondary Outcome: Serum Insulin
Description: Serum insulin measured for on day -2 and day 8 for AUEC0-5 and AUEC0-12. AUEC0-5: The area under the effect concentration-time curve over the time interval 0 to 5.
  AUEC0-12: The area under the effect concentration-time curve over the time interval 0 to 12.
Time Frame: 0.0h, 2h, 5h, 7h, 10h, 12h on day -2 & day 8
Population: PDS
Measure: Mean (Standard Deviation); unit: µU*h/mL
Arm/Group | Placebo | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9
µU*h/mL
  AUEC0-5 (12,9,9,9,9) on day-2 | 134 (52.5) | 185 (79.2) | 175 (70.7) | 137 (64.7) | 119 (35.9)
  AUEC0-12 (12,9,9,9,9) on day-2 | 300 (111) | 474 (149) | 471 (143) | 336 (161) | 282 (41.6)
  AUEC0-5 (11,9,8,9,9) on day8 | 122 (52.0) | 174 (80.9) | 180 (74.7) | 117 (103) | 101 (37.2)
  AUEC0-12 (11,9,7,9,8) on day8 | 288 (97.1) | 417 (132) | 387 (154) | 266 (193) | 275 (72.4)

21. Secondary Outcome: Serum Insulin
Description: Serum insulin measured for on day -2 and day 8 for Emax0-5, Emax0-12, Emin0-5 and Emin0-12.
  Emax: Maximum effect (maximum measured concentration of glucose or insulin in plasma) & Emin: Minimum effect (minimum measured concentration of glucose or insulin in plasma)
Time Frame: 0.0h, 2h, 5h, 7h, 10h, 12h on day -2 & day 8
Population: PDS
Measure: Mean (Standard Deviation); unit: µU/mL
Arm/Group | Placebo | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9
µU/mL
  Emax,0-5 (12,9,9,9,9) on day-2 | 38.1 (17.3) | 55.2 (29.9) | 51.2 (23.4) | 40.2 (19.4) | 35.2 (15.5)
  Emax,0-12 (12,9,9,9,9) on day-2 | 45.4 (12.6) | 68.5 (25.3) | 72.1 (27.7) | 48.7 (30.9) | 45.3 (11.3)
  Emin,0-5 (12,9,9,9,9) on day-2 | 10.3 (5.46) | 14.1 (5.45) | 13.7 (4.62) | 9.16 (7.59) | 7.86 (2.18)
  Emin,0-12 (12,9,9,9,9) on day-2 | 9.98 (4.86) | 14.1 (5.45) | 13.5 (4.37) | 9.16 (7.59) | 7.86 (2.18)
  Emax,0-5 (11,9,8,9,9) on day8 | 35.6 (15.6) | 56.0 (32.1) | 56.3 (25.4) | 36.2 (37.3) | 29.6 (11.7)
  Emax,0-12 (11,9,8,9,9) on day8 | 42.6 (13.1) | 70.2 (26.1) | 68.6 (31.1) | 44.4 (35.5) | 37.3 (8.10)
  Emin,0-5 (11,9,8,9,9) on day8 | 7.55 (3.82) | 8.63 (3.39) | 10.7 (5.60) | 5.33 (3.14) | 3.96 (2.79)
  Emin,0-12 (11,9,8,9,9) on day8 | 7.41 (3.90) | 8.53 (3.46) | 10.7 (5.60) | 5.17 (3.19) | 3.96 (2.79)

ADVERSE EVENTS:
Time Frame: day1 to day21
Arm/Group | Placebo | Empagliflozin 2.5 mg qd | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Empagliflozin 100 mg qd
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 5/12 | 6/9 | 5/9 | 5/9 | 3/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Empagliflozin 2.5 mg qd (N=9) | Empagliflozin 10 mg qd (N=9) | Empagliflozin 25 mg qd (N=9) | Empagliflozin 100 mg qd (N=9)
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Injection site thrombosis (General disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.